CLINICAL TRIAL: NCT04064983
Title: An Expanded Access IND to Evaluate the Safety and Efficacy of Autologous HB-adMSCs for the Treatment of a Single Patient With Polyneuropathy
Brief Title: Individual Patient Expanded Access IND to Treat Polyneuropathy
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBPN01
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Polyneuropathies
Keywords: Polyneuoropathy; POEMS; Pain; Stem cells; Neuropathic Pain
MeSH Terms: conditions — Polyneuropathies; Pain; Neuralgia

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: HB-adMSCs — Hope Biosciences autologous adipose-derived mesenchymal stem cells

SUMMARY:
This Individual Patient Expanded Access IND has been created as requested by an 58-year-old man who suffers from Polyneuropathy due to Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal gammopathy, and Skin abnormalities (POEMS) Syndrome. The patient will receive 8 infusions of 200 million cells every four weeks during a 28-week period to relieve the symptoms of Polyneuropathy arising due to POEMS.

DETAILED DESCRIPTION:
A screening visit will be conducted to assess the eligibility for this investigation. If the participant qualifies the expanded access program eligibility requirements, he will be treated with the investigational product in the following manner:

The patient will receive 8 infusions of 200 million cells every four weeks during a 28-week period.

This is an Individual Patient Expanded Access IND to evaluate the safety and preliminary efficacy of autologous HB-adMSCs for treating a single patient with Polyneuropathy due to POEMS Syndrome. The expanded access program will include a screening period of up to 28 days, a 28-week treatment period, a safety follow-up, and a 52-week end-of-study visit.

An informed consent form will be given to the participant, who will sign before any procedures.

The informed consent form will include information about this expanded access and all the aspects considered during this process. The following are components of the informed consent process that research personnel should adhere to:

* The principal investigator and team will make sure the participant is alert and able to read and understand the language in the consent form.
* The principal investigator and team will ensure the participant takes ample time to read the consent form carefully.
* The principal investigator and team will ensure the consent form is carefully explained to the participant or legal guardian. Any questions or concerns should be addressed before signing the document.
* Other aspects to consider, such as voluntary participation in the expanded access program, will be followed according to FDA guidance, IRB Guidelines for Researchers and Sponsor standard operating procedure

The participant is required to complete the subsequent visits after they have given their informed consent.

* Visit 1 - Screening during this period, the principal investigator will determine whether the screened participant is eligible and whether the next visit can be scheduled. Once the principal investigator has evaluated the eligibility (up to 28 days), the patient will be scheduled for the first infusion.
* Visit 2 - Infusion 1 (Baseline): this visit will be a starting point for comparing participants' data. During this visit, the patient will receive the 1st investigational product via intravenous infusion, with rigorous monitoring of vital signs for a total of 2 hours.
* Visit 3 to 9 - During these visits, the patient will receive intravenous infusions of HB-adMSCs while her vital signs are precisely monitored for a total of 2 hours.
* Follow-Up Visit - During this safety follow-up visit, the principal investigator will evaluate the safety of the investigational product by conducting several assessments described in the Schedule of Assessments table.
* End of Study - At the end of the expanded access program visit, the principal investigator will conduct various evaluations to determine the patient's physical condition and assess whether there have been any safety events resulting from the participation in the expanded access program.

ELIGIBILITY:
Inclusion Criteria

* Patient diagnosed with Polyneuropathy due to POEMS Syndrome.
* Patient must have banked his stem cells at Hope Biosciences LLC.

Exclusion Criteria

* The patient has any active infection requiring medications.
* The patient has any suicidal ideation during the screening visit.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Cheng, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States